CLINICAL TRIAL: NCT01637142
Title: An Absolute Bioavailability Study of LY2140023 and LY404039 in Healthy Subjects Using the Intravenous Tracer Method
Brief Title: A Study of LY2140023 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12682; H8Y-MC-HBCU (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2012-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — LY 2140023

ARMS (2):
- LY2140023 + [14C]-LY2140023 (Experimental): Treatment Period 1: On Day 1, a single oral dose of 80 milligrams (mg) LY2140023 (parent compound) followed by a single 2-hour intravenous (IV) infusion of approximately 100 micrograms (µg) LY2140023 containing approximately 100 nanocuries (nCi) [14C]-LY2140023.
  Interventions: Drug: LY2140023; Drug: 14C-LY2140023
- LY2140023 + [14C]-LY404039 (Experimental): Treatment Period 2: On Day 1, a single oral dose of 80 mg LY2140023 (parent compound) followed by a single 2-hour IV infusion of approximately 100 µg LY404039 containing approximately 100 nCi [14C]-LY404039 (active metabolite).
  Interventions: Drug: LY2140023; Drug: 14C-LY404039

INTERVENTIONS:
Drug: LY2140023 — Administered orally.
Drug: 14C-LY2140023 — Administered IV.
  Arms: LY2140023 + [14C]-LY2140023
Drug: 14C-LY404039 — Administered IV.
  Arms: LY2140023 + [14C]-LY404039

SUMMARY:
The purpose of this study is to assess the extent and rate of absorption of LY2140023 in healthy participants. The study has two periods. In Treatment Period 1, participants will receive a single oral dose of 80 milligrams (mg) LY2140023 followed by a 2-hour intravenous (IV) infusion of approximately 100 micrograms (µg) LY2140023 containing approximately 100 nanocuries (nCi) [14C]-LY2140023. In Treatment Period 2, participants will receive an oral dose of 80 mg LY2140023 followed by a 2-hour IV infusion of approximately 100 µg LY404039 containing approximately 100 nCi [14C]-LY404039. There will be at least a 3-day washout between doses.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females of non-childbearing potential, as determined by medical history and physical examination
* Male participants: must agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023, and agree not to donate sperm for 3 months following the last dose of LY2140023
* Female participants of non-childbearing potential i.e. postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy or confirmed tubal occlusion (not tubal ligation). Postmenopausal is defined as spontaneous amenorrhea for at least 12 months and a plasma follicle-stimulating hormone (FSH) level >40 million international units/milliliter (mIU/mL), unless the participant is taking hormone replacement therapy
* Have given written informed consent approved by Lilly and the chosen ethical review board (ERB)
* Have venous access sufficient to allow for intravenous infusion and blood sampling

Exclusion Criteria:

* Are currently enrolled in or have completed or discontinued within the last 90 days from a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated in any clinical trial involving a radiolabeled investigational product or been exposed to radiolabeled substances (for treatment or diagnosis) within the last 12 months
* Have known allergies to LY2140023 or LY404039, related compounds, or any components of the formulation
* Are persons who have previously withdrawn from this study or any other study investigating LY2140023 after receiving at least 1 dose of LY2140023
* Show evidence or any history of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* Have increased risk of seizures based on a history of:

  * One or more seizures (except for a single simple febrile seizure [lacking focality, lasting less than 15 minutes, and not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * Head trauma with loss of consciousness or a post-concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * CNS infection, uncontrolled migraine, or transient ischemic attack (TIA) within 1 year; stroke with persistent neurological deficit (focal or diffuse), uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning. TIA is defined as a "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * Brain surgery
  * Electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, or sharp-slow wave complexes, or as locally defined)
  * Brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (except hydrocephalus treated by shunt and without neurological deficit)
* Show evidence of active renal disease (for example, diabetic renal disease, polycystic kidney disease) or creatinine clearance less than 80 milliliters/minute (mL/min) as determined by the Cockroft Gault formula
* Show evidence or any history of known substance dependence or abuse at any time (according to Diagnostic and Statistical Manual of Mental Disorders [DSM-IV] diagnosis), or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a clinically significant abnormality in the neurological examination
* Participants judged prior to randomization to be at suicidal risk by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral 80 mg LY2140023 on Two Separate Occasions: Participants received a single oral dose of 80 milligrams (mg) LY2140023 (parent compound) on 2 separate occasions.
  In Treatment Period 1, a single oral dose of 80 mg LY2140023 followed by a single 2-hour intravenous (IV) infusion of approximately 100 micrograms (µg) LY2140023 containing approximately 100 nanocuries (nCi) [14C]-LY2140023.
  In Treatment Period 2, a single oral dose of 80 mg LY2140023 followed by a single 2-hour IV infusion of approximately 100 µg LY404039 (active metabolite) containing approximately 100 nCi [14C]-LY404039.
  There was a washout period of at least 3 days between Treatment Period 1 and Treatment Period 2.
Period: Treatment Period 1
Arm/Group | Oral 80 mg LY2140023 on Two Separate Occasions
Started | 18
Received at Least 1 Dose of Study Drug | 18
Completed | 18
Not Completed | 0
Period: Washout Period (at Least 3 Days)
Arm/Group | Oral 80 mg LY2140023 on Two Separate Occasions
Started | 18
Completed | 17
Not Completed | 1
Not completed — Physician Decision | 1
Period: Treatment Period 2
Arm/Group | Oral 80 mg LY2140023 on Two Separate Occasions
Started | 17
Received at Least 1 Dose of Study Drug | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at last 1 dose of LY2140023.
Groups:
- Oral 80 mg LY2140023 on Two Separate Occasions: Participants received a single oral dose of 80 mg LY2140023 (parent compound) on 2 separate occasions.
  In Treatment Period 1, a single oral dose of 80 mg LY2140023 followed by a single 2-hour IV infusion of approximately 100 µg LY2140023 containing approximately 100 nCi [14C]-LY2140023.
  In Treatment Period 2, a single oral dose of 80 mg LY2140023 followed by a single 2-hour IV infusion of approximately 100 µg LY404039 (active metabolite) containing approximately 100 nCi [14C]-LY404039.
  There was a washout period of at least 3 days between Treatment Period 1 and Treatment Period 2.
Arm/Group | Oral 80 mg LY2140023 on Two Separate Occasions
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY2140023 and LY404039 in Treatment Period 1
Description: Exposure of LY2140023 (parent compound), LY404039 (active metabolite), 14C-radiolabeled LY2140023, and 14C-radiolabeled LY404039 in terms of Area Under the Concentration Versus Time Curve from time 0 extrapolated to infinity (AUC[0-inf]) is summarized for participants in Treatment Period 1.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 12, 16 and 24 hours postdose
Population: Participants who received oral LY2140023 with IV [14C]-LY2140023 and had evaluable pharmacokinetic (PK) concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours per milliliter
Groups:
- Oral 80 mg LY2140023 and IV LY2140023/[14C]-LY2140023: In Treatment Period 1, a single oral dose of 80 mg LY2140023 followed by a single 2-hour IV infusion of approximately 100 µg LY2140023 containing approximately 100 nCi [14C]-LY2140023.
Arm/Group | Oral 80 mg LY2140023 and IV LY2140023/[14C]-LY2140023
Number analyzed (Participants) | 18
nanograms times hours per milliliter
  LY2140023 (parent compound) | 1160 (28)
  LY404039 (active metabolite) | 2620 (23)
  [14C]-LY2140023 (parent) | 2.01 (22)
  [14C]-LY404039 (active metabolite) | 6.19 (20)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY2140023 and LY404039 in Treatment Period 2
Description: Exposure of LY2140023 (parent compound), LY404039 (active metabolite), and 14C-radiolabeled LY404039 in terms of Area Under the Concentration Versus Time Curve from time 0 extrapolated to infinity (AUC[0-inf]) is summarized for participants in Treatment Period 2.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16 and 24 hours postdose
Population: Participants who received oral LY2140023 with IV [14C]-LY404039 and had evaluable PK concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours per milliliter
Groups:
- Oral 80 mg LY2140023 and IV LY404039/[14C]-LY404039: In Treatment Period 2, a single oral dose of 80 mg LY2140023 (parent compound) followed by a single 2-hour IV infusion of approximately 100 µg LY404039 (active metabolite) containing approximately 100 nCi [14C]-LY404039.
Arm/Group | Oral 80 mg LY2140023 and IV LY404039/[14C]-LY404039
Number analyzed (Participants) | 17
nanograms times hours per milliliter
  LY2140023 (parent compound) | 1200 (27)
  LY404039 (active metabolite) | 2690 (21)
  [14C]-LY404039 (active metabolite) | 7.69 (20)

ADVERSE EVENTS:
Groups:
- Oral 80 mg LY2140023 and IV LY2140023/[14C]-LY2140023: Treatment Period 1: On Day 1, a single oral dose of 80 mg LY2140023 (parent compound) followed by a single 2-hour IV infusion of approximately 100 µg LY2140023 containing approximately 100 nCi [14C]-LY2140023.
- Oral 80 mg LY2140023 and IV LY404039/[14C]-LY404039: Treatment Period 2: On Day 1, a single oral dose of 80 mg LY2140023 (parent compound) followed by a single 2-hour IV infusion of approximately 100 µg LY404039 (active metabolite) containing approximately 100 nCi [14C]-LY404039.
Arm/Group | Oral 80 mg LY2140023 and IV LY2140023/[14C]-LY2140023 | Oral 80 mg LY2140023 and IV LY404039/[14C]-LY404039
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 8/18 | 10/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral 80 mg LY2140023 and IV LY2140023/[14C]-LY2140023 (N=18) | Oral 80 mg LY2140023 and IV LY404039/[14C]-LY404039 (N=17)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 2 (2)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days